CLINICAL TRIAL: NCT03494127
Title: Development of Advanced Personalized Modular Pressure Relief Seating Cushion Systems: Testing and User Evaluation
Brief Title: User Evaluation of Advanced Personalized Modular Pressure Relief Seating Cushion Systems
Acronym: Squishycushion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: A2434-R; I01RX002434 (NIH)
Record Dates: First submitted 2018-03-27; First posted 2018-04-11 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Mobility Impairment
Keywords: wheelchair seating; tissue health

STUDY DESIGN:
Intervention Model Description: Repeated measures crossover clinical study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): DAILY COMMUNITY USE OF GEL BALL FITTED MODULAR CUSHION for 2 weeks followed by DAILY COMMUNITY USE OF SQUISHINS FITTED MODULAR CUSHION for 2 weeks
  Interventions: Device: Use of GEL BALL FITTED MODULAR CUSHION; Device: Use of SQUISHINS FITTED MODULAR CUSHION
- Group B (Experimental): DAILY COMMUNITY USE OF SQUISHINS FITTED MODULAR CUSHION for 2 weeks followed by DAILY COMMUNITY USE OF GEL BALL FITTED MODULAR CUSHION for 2 weeks
  Interventions: Device: Use of GEL BALL FITTED MODULAR CUSHION; Device: Use of SQUISHINS FITTED MODULAR CUSHION

INTERVENTIONS:
Device: Use of GEL BALL FITTED MODULAR CUSHION — DAILY COMMUNITY USE OF GEL BALL FITTED MODULAR CUSHION for 2 weeks
Device: Use of SQUISHINS FITTED MODULAR CUSHION — DAILY COMMUNITY USE OF SQUISHINS FITTED MODULAR CUSHION for 2 weeks

SUMMARY:
30 Veterans who are full-time wheelchair users will use personalized modular cushions for two weeks each. Personalized cushions will be created using a cushion fitting process the investigators have already developed and tested. Microenvironmental conditions will be monitored during use. A cost analysis will ensure the customized modular cushion applies value-driven principles. User satisfaction will be measured along with the effects on daily function, skin status and seated tissue health.

DETAILED DESCRIPTION:
A repeated measures clinical study design will be carried out with 30 Veterans. 'Pre-baseline' seated interface pressures will be assessed with study participants sitting on their own cushions and pelvic region skin checks carried out by the study Research Nurse. All participants will then receive customized modular cushions. Participants will be randomly assigned to Group A or Group B using a modified randomization scheme. Group A participants will first use a gel ball fitted cushion for 2 weeks during all daily living activities while seated in their wheelchair followed by use of a SquishINS fitted cushion for 2 weeks. Group B will first use the SquishINS fitted cushion then a gel ball fitted cushion. Seated interface pressure distribution will be obtained at the beginning and end of each test period. A dual temperature and humidity sensor placed in the cushion will enable continuous monitoring of microenvironmental status during use. The study Research Nurse will repeat the pelvic region skin check and participants will complete a questionnaire based on the QUEST 2.0 user satisfaction instrument. All responses will be documented as part of the QS/DC program.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with mobility impairments requiring full time use of a power or manual wheelchair who are served through the LSCDVAMC Wheeled Mobility Clinic.

Exclusion Criteria:

* Pregnancy
* Inability to remain seated in the wheelchair for more than 4 hours/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-08-23 (Estimated); Primary Completion 2027-12-28 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Seated interface pressure distribution | After each 2 week period of cushion use for 5 minutes at each assessment
  Interface pressure distribution (mmHg) will be recorded using the Tekscan CONFORMat® Pressure Measurement System. Real-time 3-D images of pressure distribution at the seating interface are produced using graphical display software.
Microenvironmental status I - temperature | Continuously during each 2 week period of cushion use
  A dual temperature and humidity sensor will be placed in the cushion for continuous monitoring of microenvironmental status. At the end of each test period, microenvironmental temperature status data (deg C) will be downloaded for analysis.
Microenvironmental status II - humidity | Continuously during each 2 week period of cushion use
  A dual temperature and humidity sensor will be placed in the cushion for continuous monitoring of microenvironmental status. At the end of each test period, microenvironmental humidity status data (relative humidity units) will be downloaded for analysis.

SECONDARY OUTCOMES:
User satisfaction questionnaire | After each 2 week period of cushion use for 5 minutes at each assessment
  Questionnaire based on the QUEST 2.0 user satisfaction instrument

OTHER OUTCOMES:
Skin health checks | Before and after cushion use (2 week period)
  Pelvic region skin checks will be carried out by the study Research Nurse to ensure there are no areas of redness or breakdown.

CONTACTS AND LOCATIONS:
Overall Officials: Kath M. Bogie, PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No